CLINICAL TRIAL: NCT00605072
Title: The Antihypertensives and Vascular, Endothelial and Cognitive Function Trial (AVEC Trial)
Brief Title: The Antihypertensives and Vascular, Endothelial and Cognitive Function Trial
Acronym: AVEC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Ihab Hajjar, Assistant Professor of Medicine, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0127; K23AG030057 (NIH)
Record Dates: First submitted 2008-01-11; First posted 2008-01-30 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-01

CONDITIONS: Cognitive Impairment; Hypertension; Aging
Keywords: cognitive disorders; angiotensin receptor blockers
MeSH Terms: conditions — Cognitive Dysfunction; Hypertension | interventions — candesartan; candesartan cilexetil; Lisinopril; Hydrochlorothiazide; Nifedipine; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Candesartan (Experimental): Angiotensin Receptor Blocker
  Interventions: Drug: candesartan; Drug: nifedipine, long acting; Drug: metoprolol, long-acting
- Lisinopril (Experimental): Angiotensin-Converting Enzyme (ACE) Inhibitor
  Interventions: Drug: lisinopril; Drug: nifedipine, long acting; Drug: metoprolol, long-acting
- HCTZ (Active Comparator): Hydrochlorothiazide (diuretic)
  Interventions: Drug: hydrochlorothiazide

INTERVENTIONS:
Drug: candesartan — orally 8 mg increased to 16 mg then 32 mg to achieve target blood pressure of 140/90, then daily for 12 months
  Other Names: Atacand
  Arms: Candesartan
Drug: lisinopril — orally 10 mg increased to 20 mg then 40 mg to achieve target blood pressure of 140/90, then daily for 12 months
  Other Names: Prinivil
  Arms: Lisinopril
Drug: hydrochlorothiazide — orally 12.5 mg increased to 25 mg to achieve target blood pressure of 140/90, then daily for 12 months
  Other Names: HCTZ, multiple brand names
  Arms: HCTZ
Drug: nifedipine, long acting — If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 30 mg increased to 60 mg and 90 mg in 2 week increments
  Other Names: Procardia XL
  Arms: Candesartan; Lisinopril
Drug: metoprolol, long-acting — If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 12.5 mg increased to 25 mg and 50 mg
  Other Names: Lopressor, Toprol XL
  Arms: Candesartan; Lisinopril

SUMMARY:
The purpose of this study is to examine the effects of blood pressure medications on cognition and blood flow in hypertensive elderly patients with cognitive impairment. The hypothesis is that treatment with an angiotensin receptor blocker (ARB) or an angiotensin-converting enzyme inhibitor (ACEI) will be associated with a slower rate of further cognitive decline, improved cerebral blood flow and its regulation, and preserved physical function as compared to treatment with a diuretic (HCTZ), independent of blood pressure level.

DETAILED DESCRIPTION:
There is mounting evidence that hypertension, which affects more than 65% of the US elderly population, accelerates cognitive decline and increases the risk of functional disability among older individuals. Hypertension is also associated with cerebral blood flow reduction and dysregulation which contribute to further cognitive and functional impairment. Drugs that inhibit angiotensin II (ACEI and ARB) are commonly used antihypertensives and may have a protective effect on cognitive function, cerebral blood flow and physical function compared to other antihypertensives such as hydrochlorothiazide (HCTZ).

A total of 100 individuals will be recruited for this pilot 3-arm randomized study to investigate the effects of: (i) 12 months treatment with candesartan (ARB) compared to hydrochlorothiazide (HCTZ) and (ii) 12 months treatment with lisinopril (ACEI) compared to HCTZ and (iii) to estimate the effect size difference between lisinopril and losartan on cognition, cerebral blood flow regulation, and functional measures in a sample of elderly hypertensive individuals with objective evidence of cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older
* Hypertension
* Cognitive criteria: score either 10 or less out of 15 for the executive clock draw test 1 (CLOX1) or less than or equal to 1 standard deviation from the corresponding age specific mean on the immediate memory subtest

Exclusion Criteria:

* Intolerance to ACEI or ARB
* History of congestive heart failure
* History of diabetes mellitus
* History of stroke (less than 6 months)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ihab Hajjar, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - Hebrew SeniorLife, Boston, Massachusetts

REFERENCES:
- [Background] Lipsitz LA, Gagnon M, Vyas M, Iloputaife I, Kiely DK, Sorond F, Serrador J, Cheng DM, Babikian V, Cupples LA. Antihypertensive therapy increases cerebral blood flow and carotid distensibility in hypertensive elderly subjects. Hypertension. 2005 Feb;45(2):216-21. doi: 10.1161/01.HYP.0000153094.09615.11. Epub 2005 Jan 17. PMID 15655124
- [Background] Hajjar I, Hart M, Milberg W, Novak V, Lipsitz L. The rationale and design of the antihypertensives and vascular, endothelial, and cognitive function (AVEC) trial in elderly hypertensives with early cognitive impairment: role of the renin angiotensin system inhibition. BMC Geriatr. 2009 Nov 18;9:48. doi: 10.1186/1471-2318-9-48. PMID 19922631
- [Result] Hajjar I, Hart M, Chen YL, Mack W, Milberg W, Chui H, Lipsitz L. Effect of antihypertensive therapy on cognitive function in early executive cognitive impairment: a double-blind randomized clinical trial. Arch Intern Med. 2012 Mar 12;172(5):442-4. doi: 10.1001/archinternmed.2011.1391. No abstract available. PMID 22412114
- [Derived] Hajjar I, Hart M, Chen YL, Mack W, Novak V, C Chui H, Lipsitz L. Antihypertensive therapy and cerebral hemodynamics in executive mild cognitive impairment: results of a pilot randomized clinical trial. J Am Geriatr Soc. 2013 Feb;61(2):194-201. doi: 10.1111/jgs.12100. Epub 2013 Jan 25. PMID 23350899

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisinopril: Angiotensin-Converting Enzyme (ACE) Inhibitor: lisinopril : orally 10 mg increased to 20 mg then 40 mg to achieve target blood pressure of 140/90, then daily for 12 months
  nifedipine, long acting : If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 30 mg increased to 60 mg and 90 mg in 2 week increments
  metoprolol, long-acting : If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 12.5 mg increased to 25 mg and 50 mg
- Candesartan: Angiotensin Receptor Blocker: candesartan : orally 8 mg increased to 16 mg then 32 mg to achieve target blood pressure of 140/90, then daily for 12 months
  nifedipine, long acting : If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 30 mg increased to 60 mg and 90 mg in 2 week increments
  metoprolol, long-acting : If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 12.5 mg increased to 25 mg and 50 mg
- HCTZ: hydrochlorothiazide : orally 12.5 mg increased to 25 mg to achieve target blood pressure of 140/90, then daily for 12 months
  nifedipine, long acting : If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 30 mg increased to 60 mg and 90 mg in 2 week increments
  metoprolol, long-acting : If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 12.5 mg increased to 25 mg and 50 mg
Period: Overall Study
Arm/Group | Lisinopril | Candesartan | HCTZ
Started | 18 | 20 | 15
Completed | 11 | 9 | 11
Not Completed | 7 | 11 | 4

BASELINE CHARACTERISTICS:
Groups:
- ACEI (Lisinopril): Angiotensin-Converting Enzyme (ACE) Inhibitor: lisinopril : orally 10 mg increased to 20 mg then 40 mg to achieve target blood pressure of 140/90, then daily for 12 months
  nifedipine, long acting : If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 30 mg increased to 60 mg and 90 mg in 2 week increments
  metoprolol, long-acting : If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 12.5 mg increased to 25 mg and 50 mg
- ARB (Candesartan): Angiotensin Receptor Blocker: candesartan : orally 8 mg increased to 16 mg then 32 mg to achieve target blood pressure of 140/90, then daily for 12 months
  nifedipine, long acting : If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 30 mg increased to 60 mg and 90 mg in 2 week increments
  metoprolol, long-acting : If needed to achieve target blood pressure of 140/90, added to ARB or ACEI at 12.5 mg increased to 25 mg and 50 mg
- Total: Total of all reporting groups
Arm/Group | ACEI (Lisinopril) | ARB (Candesartan) | HCTZ | Total
Number analyzed (Participants) | 18 | 20 | 15 | 53
Age Continuous [Mean (Standard Deviation); unit: years] | 71 (7) | 71 (9) | 71 (7) | 71 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 9 | 31
  Male | 7 | 9 | 6 | 22
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 15 | 53

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Assessment: Trail Making Test Part B
Description: This test requires the connection of sequentially numbered circles (A), and the connection of circles marked by numbers and letters in alternating sequence (B). This test is considered a benchmark of executive function. The test score is the time required to complete the task in seconds.
Time Frame: Baseline-12 months
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | ACEI (Lisinopril) | ARB (Candesartan) | HCTZ
Number analyzed (Participants) | 18 | 20 | 15
seconds | -14 (9) | 17 (10) | 4 (9)
Statistical Analysis 1: Comparison: ACEI (Lisinopril) vs ARB (Candesartan) vs HCTZ; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — p-value for between group comparison (group*visit); Adjusted for baseline AGE and Mini-Mental-State-Examination

2. Secondary Outcome: Blood Pressure Outcome: Systolic BP
Description: Blood pressure was measured as follows: the participant was in the sitting position, rested for 5 minutes, no caffeine or smoking 2 hours prior to measurement, using appropriate cuff size (covering 60% of upper arm length and 80% of arm circumference), correct cuff placement (1-2 inches above brachial pulse on bare arm), and the bell of the stethoscope. The systolic blood pressure was defined as the pressure corresponding to the first korotkoff sounds (K1) and the diastolic as the pressure corresponding to the last korotkoff sound (K5). Blood pressure was measured in both arms and recorded
Time Frame: Baseline-12 months
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | ACEI (Lisinopril) | ARB (Candesartan) | HCTZ
Number analyzed (Participants) | 17 | 17 | 13
mm Hg | 28 (5) | 27 (5) | 21 (5)
Statistical Analysis 1: Comparison: ACEI (Lisinopril) vs ARB (Candesartan) vs HCTZ; Test type: Superiority or Other; p = 0.74, Mixed Models Analysis; adjusted for age

3. Secondary Outcome: Blood Flow Velocity, Sitting
Description: This reports the change in the least square mean from baseline to 12 months, adjusted for age
Time Frame: Baseline-12 months
Measure: Least Squares Mean (Standard Error); unit: cm/sec
Arm/Group | ACEI (Lisinopril) | ARB (Candesartan) | HCTZ
Number analyzed (Participants) | 17 | 17 | 13
cm/sec | -0.3 (1.5) | -2.85 (1.71) | 0.35 (1.68)
Statistical Analysis 1: Comparison: ACEI (Lisinopril) vs ARB (Candesartan) vs HCTZ; Test type: Superiority or Other; p = 0.81, Mixed Models Analysis; Adjusted for age at baseline

4. Primary Outcome: Cognitive Assessment: Hopkins Verbal Learning- Immediate Recall
Description: This is a 12-item list learning test in which individuals are presented three learning and recall trials followed by a delayed recall and 24 item recognition test. The HVLT-R has been identified as an ideal memory measure for elderly patients, and appropriate reliability and validity have been shown in older individuals. The test score is the number of correct answers in the delayed recall ( score range 0-12)
Time Frame: Baseline-12 months
Measure: Least Squares Mean (Standard Error); unit: number words remembered
Arm/Group | ACEI (Lisinopril) | ARB (Candesartan) | HCTZ
Number analyzed (Participants) | 18 | 20 | 15
number words remembered | -1 (1) | -2 (1) | -3 (1)
Statistical Analysis 1: Comparison: ACEI (Lisinopril) vs ARB (Candesartan) vs HCTZ; Test type: Superiority or Other; p = 0.87, Mixed Models Analysis

5. Primary Outcome: Cognitive Assessment: Forward Digit Span Test
Description: This test consists of series of digits of increasing length, some of which are recited as presented, and some of which are to be recited in reversed order. The forward digit span score ranges from 0 (ie cannot repeat two digits) to 8 ( participant can repeat up to 8 digits)
Time Frame: Baseline-12 months
Measure: Least Squares Mean (Standard Error); unit: number of digits repeated
Arm/Group | ACEI (Lisinopril) | ARB (Candesartan) | HCTZ
Number analyzed (Participants) | 18 | 20 | 15
number of digits repeated | -0.3 (0.3) | 0.02 (0.04) | -0.04 (0.29)
Statistical Analysis 1: Comparison: ACEI (Lisinopril) vs ARB (Candesartan) vs HCTZ; Test type: Superiority or Other; p = 0.79, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | ACEI (Lisinopril) | ARB (Candesartan) | HCTZ
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20 | 0/15
Other Adverse Events (participants affected / at risk) | 5/18 | 6/20 | 6/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACEI (Lisinopril) (N=18) | ARB (Candesartan) (N=20) | HCTZ (N=15)
Dizziness (Nervous system disorders) | 5 | 6 | 6
Weakness or Fatigue (Nervous system disorders) | 3 | 1 | 1
Fall, non-injurious (Nervous system disorders) | 4 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 3
Hospitalization (non-elective) (Injury, poisoning and procedural complications) | 4 | 3 | 3

LIMITATIONS AND CAVEATS:
The main limitation is the small sample size. The validity of TCD measurements as an index of cerebral blood flow is based on the assumption that cerebral vessel diameters are constant but we didn't have brain imaging to validate this assumption.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No